CLINICAL TRIAL: NCT00604656
Title: A Six Months, Multi-centre, Open, Randomised, Parallel Safety and Efficacy Comparison of NovoRapid® Produced by the Current Process and Insulin Aspart With the Same Formulation as NovoRapid®, Produced by the NN2000 Process in Subjects With Type 1 Diabetes on a Basal/Bolus Regimen
Brief Title: Comparison of Insulin Aspart Produced by the NN2000 Process to the Current Process in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2000-1542
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the safety and efficacy of insulin aspart produced by current process compared to that of insulin aspart produced by NN2000 process in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 1 diabetes
* Duration of diabetes for at least 12 months
* Treatment with insulin aspart for at least 3 months before trial start
* Body Mass Index (BMI) below 35.0 kg/m2
* HbA1c below 12.0%

Exclusion Criteria:

* Total insulin dosage more than 1.4 IU/kg/day
* Recurrent major hypoglycaemia that may interfere with trial participation (as judged by the investigator)
* Known hypoglycaemia unawareness as judged by the investigator
* Known hypersensitivity or allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2003-05-05 (Actual); Primary Completion 2004-01-29 (Actual); Study Completion 2004-01-29 (Actual)

PRIMARY OUTCOMES:
Insulin aspart antibodies | After 6 months treatment

SECONDARY OUTCOMES:
Occurrence of adverse events
Incidence of hypoglycaemic episodes
HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (33):
- Czechia (2):
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Prague
- Germany (15):
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Bad Neuenahr-Ahrweiler
  - Novo Nordisk Investigational Site, Diez
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Karlsruhe
  - Novo Nordisk Investigational Site, Marktheidenfeld
  - Novo Nordisk Investigational Site, Marl
  - Novo Nordisk Investigational Site, Oberursel
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saarbrücken
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Simmern
  - Novo Nordisk Investigational Site, Speyer
  - Novo Nordisk Investigational Site, Würzburg
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Nyíregyháza
- Italy (9):
  - Novo Nordisk Investigational Site, Cagliari
  - Novo Nordisk Investigational Site, Chiavari
  - Novo Nordisk Investigational Site, Città di Castello
  - Novo Nordisk Investigational Site, Lucca
  - Novo Nordisk Investigational Site, Orvieto
  - Novo Nordisk Investigational Site, Parma
  - Novo Nordisk Investigational Site, Perugia
  - Novo Nordisk Investigational Site, Rimini
  - Novo Nordisk Investigational Site, Roma
- Poland (5):
  - Novo Nordisk Investigational Site, Bytom
  - Novo Nordisk Investigational Site, Mazowieckie
  - Novo Nordisk Investigational Site, Radom
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com